CLINICAL TRIAL: NCT05126199
Title: The Effect of Time-restricted Eating on Insulin Levels and Other Metabolic Abnormalities in Polycystic Ovarian Syndrome: A Randomised Feasibility Study of Real-world Clinical Advice
Brief Title: Time-restricted Eating to Improve Metabolic Abnormalities in Polycystic Ovarian Syndrome
Acronym: TimeMAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruairí Floyd (Other)
Collaborators: Tallaght University Hospital (Other)
Responsible Party: Sponsor-Investigator, Ruairí Floyd, Study Co-ordinator and Researcher, Tallaght University Hospital
Organization: Tallaght University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TimeMAP
Record Dates: First submitted 2021-10-28; First posted 2021-11-18 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: PCOS; Hyperinsulinemia; Insulin Resistance
Keywords: PCOS; Intermittent Fasting; Fasting; Hyperinsulinemia; Insulin Resistance
MeSH Terms: conditions — Hyperinsulinism; Insulin Resistance; Intermittent Fasting; Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted eating (Experimental): Time-restricted eating using 18:6 protocol (12 weeks)
  Washout Period (4 weeks)
  Crossover to Normal ad libitum diet (12 weeks)
  Interventions: Other: Time restricted eating
- Normal ad libitum diet (Active Comparator): Normal ad libitum dietary patterns without defined eating window, fasting or restrictions on types of food or drink consumed (12 weeks)
  Washout Period (4 weeks)
  Crossover to time-restricted eating using 18:6 protocol (12 weeks)
  Interventions: Other: Normal ad libitum diet

INTERVENTIONS:
Other: Time restricted eating — Following a 3 day baseline dietary assessment using the Nutritics 'app', patients will immediately commence time-restricted eating on a 18:6 basis (18 hours fasting, 6 hours eating window) for 12 weeks.
  Participants will consume all their meals within a daily 6-hour period of their choosing, and this may change according to patient's lifestyle and preference to reflect a real-world situation. Participants may eat ad libitum / according to appetite during the eating period. Participants will fast for 18 hours per day, consuming only plain water, unflavoured/unsweetened sparkling water, black breakfast tea or black coffee. Alcohol must not be consumed during fasting periods
  Dietary intake will again be measured using the Nutritics 'app' midpoint through the 12-week period (week 6 +/- 1 week) and in the last week of the intervention (week 11/12).
  Arms: Time restricted eating
Other: Normal ad libitum diet — Following a 3-day baseline dietary assessment using the Nutritics 'app', participants with be directed to continue with their usual dietary intake without any time-related restrictions for 12 weeks. There will be no defined eating window and fasting or restrictions regarding types of food or drink consumed.
  Dietary intake will again be measured using the Nutritics 'app' midpoint through the 12-week period (week 6 +/- 1 week) and in the last week of the intervention (week 11/12).
  Arms: Normal ad libitum diet

SUMMARY:
Polycystic ovarian syndrome (PCOS) is associated with metabolic symptoms such as hyperinsulinemia. Time-restricted eating may reduce serum insulin and improve insulin resistance in patients with PCOS. Currently, there are few studies investigating time-restricted eating in patients with PCOS. The investigators plan to test the feasibility of time-restricted eating in the management of PCOS by means of a real-world clinical intervention. The investigators will determine if an 18:6 eating protocol reduces insulin levels by means of a randomised controlled crossover trial.

DETAILED DESCRIPTION:
Background: Polycystic ovarian syndrome (PCOS) is the most common reproductive endocrinopathy in women of reproductive age with many associated metabolic symptoms, in particular hyperinsulinemia, insulin resistance and a high lifetime risk of type 2 diabetes mellitus. The effects of time-restricted eating on metabolic profiles have been investigated in many endocrinopathies, but there are minimal data in PCOS.

Methods: This study will investigate the feasibility of time-restricted eating in the management of PCOS, and its effects on insulin levels and other metabolic parameters.

To achieve this, the investigators will recruit 20 patients with PCOS (normal weight, overweight, obese).

In a randomised cross-over design, participants will be observed for two consecutive 12 week periods (with a 4 weeks washout period in between) following either 'time-restricted eating' or 'usual eating', detailed below.

1. 18:6 protocol: 18 hours of fasting and a 6-hours eating window, with no other specific dietary advice. Participants choose their own 6-hour period according to their lifestyle and preference.
2. Usual eating: follow usual eating patterns, no time restriction, no other dietary advice

When fasting, participants are permitted to consume plain water, unflavoured/unsweetened sparkling water, black breakfast tea and black coffee.

Dietary intake will be determined at baseline, at midpoint of each study arm, and at the end of the study using Nutritics software. Participants will self-record dietary intake using the Nutritics 'app'.

The primary endpoints will be serum insulin and feasibility of the intervention as well as safety, acceptability, and compliance with time-restricted eating.

Secondary endpoints will be insulin resistance (Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)), androgens (testosterone, free testosterone, dehydroepiandrosterone sulfate (DHEA-S), androstenedione, 17-Hydroxyprogesterone (17-OHP) and sex hormone binding globulin (SHBG)), appetite (10-point visual analogue scale), hunger/satiety (glucagon-like peptide 1 (GLP-1), grehlin, PYY and oxyntomodulin, fasting glucose, HbA1c, lipid profile, lipoprotein lipid A, apolipoprotein A1, apolipoprotein B, anthropometrics (weight, body mass index, hip and waist circumference), dietary intake (calorie and macronutrient intake; micronutrient intake including iron, calcium; dietary pattern including timing).

Results: Safety and acceptability will be measured by adverse event reporting and measurement of adherence. Paired t-test will be used to assess between baseline and post intervention measurements. Results considered statistically significant if p<0.05.

Discussion: Time-restricted eating has potential to aid in improvement of insulin resistance in patients with PCOS based on studies in other populations. There is no substantial literature on this subject to date in the PCOS patient cohort, with this being the first randomised study to date. The investigators will discuss the effects of time-restricted eating on insulin levels in the specific population of women with PCOS based on the results.

ELIGIBILITY:
Inclusion Criteria:

* Adult women of reproductive age with confirmed diagnosis of PCOS (Rotterdam Criteria, including at least 2 of 3 characteristics: oligomenorrhea, clinical and/or biochemical hyperandrogenism and ultrasound criteria)
* No BMI restriction
* Able and willing to provide explicit, informed consent

Exclusion Criteria:

* Type 1 diabetes, medication-controlled type 2 diabetes
* Pregnancy
* Currently participating in weight loss programme, or reported weight change in last 3 months (>5% of current body weight)
* Documented history of eating disorder
* Ovulation medication, such as clomiphene citrate
* Weight loss medication affecting weight or appetite in last 6 months, including weight loss medications, antipsychotic drugs or other medications as determine by the physician (eg. Semaglutide, liraglutide, orlistat, amphetamines, Qsymia (phentermine-topiramate), bupropion-naltrexone (Contrave))
* Known liver, renal or thyroid dysfunction (not including non-alcoholic fatty liver disease with hypothyroidism on treatment or subclinical hypothyroidism seen in a large proportion of patients with PCOS)
* Unable to participate in follow-up for at least 24 weeks
* Unable or unwilling to provide explicit, informed consent

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Drop-out rate | 6 weeks
  Assessing intervention feasibility
Drop-out rate | 12 weeks
  Assessing intervention feasibility
Adverse outcomes as assessed by CTCAE v4.0 | 6 weeks
  Assessing intervention feasibility
Adverse outcomes as assessed by CTCAE v4.0 | 12 weeks
  Assessing intervention feasibility
Change in serum insulin | 6 weeks
  Measured with serum insulin levels to assess effects
Change in serum insulin | 12 weeks
  Measured with serum insulin levels to assess effects
Change in food diaries | 6 weeks
  Assessment of change of eating behaviours
Change in food diaries | 12 weeks
  Assessment of change of eating behaviours

SECONDARY OUTCOMES:
Change in insulin resistance | 6 weeks
  Assessed by Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) and other ratio calculations measuring insulin resistance
Change in insulin resistance | 12 weeks
  Assessed by Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) and other ratio calculations measuring insulin resistance
Change in testosterone levels | 6 weeks
  Assessed by plasma testosterone
Change in testosterone levels | 12 weeks
  Assessed by plasma testosterone
Change in free testosterone levels | 6 weeks
  Assessed by plasma free testosterone
Change in free testosterone levels | 12 weeks
  Assessed by plasma free testosterone
Change in dehydroepiandrosterone sulfate (DHEA-S) levels | 6 weeks
  Assessed by plasma dehydroepiandrosterone sulfate (DHEA-S)
Change in dehydroepiandrosterone sulfate (DHEA-S) levels | 12 weeks
  Assessed by plasma dehydroepiandrosterone sulfate (DHEA-S)
Change in androstenedione levels | 6 weeks
  Assessed by plasma androstenedione
Change in androstenedione levels | 12 weeks
  Assessed by plasma androstenedione
Change in sex hormone binding globulin (SHBG) levels | 6 weeks
  Assessed by plasma sex hormone binding globulin (SHBG)
Change in sex hormone binding globulin (SHBG) levels | 12 weeks
  Assessed by plasma sex hormone binding globulin (SHBG))
Change in 17-Hydroxyprogesterone (17-OHP) levels | 6 weeks
  Assessed by 17-Hydroxyprogesterone (17-OHP)
Change in 17-Hydroxyprogesterone (17-OHP) levels | 12 weeks
  Assessed by 17-Hydroxyprogesterone (17-OHP)
Change in appetite | 6 weeks
  Measured by a validated 10-point visual analogue scale on a scale of 1-10, 1 being not hungry at all and 10 being very hungry
Change in appetite | 12 weeks
  Measured by a validated 10-point visual analogue scale on a scale of 1-10, 1 being not hungry at all and 10 being very hungry
Change in markers of satiety | 6 weeks
  Assess by plasma GLP-1
Change in markers of satiety | 12 weeks
  Assess by plasma GLP-1
Change in markers of satiety | 6 weeks
  Assess by plasma PYY
Change in markers of satiety | 12 weeks
  Assess by plasma PYY
Change in markers of satiety | 6 weeks
  Assess by plasma oxyntomodulin
Change in markers of satiety | 12 weeks
  Assess by plasma oxyntomodulin
Change in markers of hunger | 6 weeks
  Assess by plasma ghrelin
Change in markers of hunger | 12 weeks
  Assess by plasma ghrelin
Change in fasting glucose | 6 weeks
  Assessed in serum glucose measurements
Change in fasting glucose | 12 weeks
  Assessed in serum glucose measurements
Change in HbA1c | 6 weeks
  Assessed in serum HbA1c measurements
Change in HbA1c | 12 weeks
  Assessed in serum HbA1c measurements
Change in lipids | 6 weeks
  Assessed by Lipid profile
Change in lipids | 12 weeks
  Assessed by Lipid profile
Change in lipids | 6 weeks
  Assessed by Lipoprotein lipid A levels
Change in lipids | 12 weeks
  Assessed by Lipoprotein lipid A levels
Change in lipids | 6 weeks
  Assessed by Apolipoprotein A1 levels
Change in lipids | 12 weeks
  Assessed by Apolipoprotein A1 levels
Change in lipids | 6 weeks
  Assessed by Apolipoprotein B levels
Change in lipids | 12 weeks
  Assessed by Apolipoprotein B levels
Change in body weight | 6 weeks
  Body weight (kg)
Change in body weight | 12 weeks
  Body weight (kg)
Change in body mass index | 6 weeks
  BMI (kg/m2)
Change in body mass index | 12 weeks
  BMI (kg/m2)
Change in anthropometric measurements (waist circumference) | 6 weeks
  Waist circumference (cm)
Change in anthropometric measurements (waist circumference) | 12 weeks
  Waist circumference (cm)
Change in anthropometric measurements (waist-hip ratio) | 6 weeks
  Waist-hip ratio
Change in anthropometric measurements (waist-hip ratio) | 12 weeks
  Waist-hip ratio
Change in dietary intake | 6 weeks
  Assessed using interval dietary assessments with Nutritics 'app'
Change in dietary intake | 12 weeks
  Assessed using interval dietary assessments with Nutritics 'app'

CONTACTS AND LOCATIONS:
Overall Officials: Lucy-Ann Behan, MD, Principal Investigator — Robert Graves Institute of Endocrinology, Tallaght University Hospital; Sinead Duggan, R.D. PhD, Study Director — University of Dublin, Trinity College
Locations (1):
- Robert Graves Institute of Endocrinology, Tallaght University Hospital, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asemi Z, Samimi M, Taghizadeh M, Esmaillzadeh A. Effects of Ramadan Fasting on Glucose Homeostasis, Lipid Profiles, Inflammation and Oxidative Stress in Women with Polycystic Ovary Syndrome in Kashan, Iran. Arch Iran Med. 2015 Dec;18(12):806-10. PMID 26621011
- [Background] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Fertil Steril. 2018 Aug;110(3):364-379. doi: 10.1016/j.fertnstert.2018.05.004. Epub 2018 Jul 19. PMID 30033227
- [Background] Anton SD, Moehl K, Donahoo WT, Marosi K, Lee SA, Mainous AG 3rd, Leeuwenburgh C, Mattson MP. Flipping the Metabolic Switch: Understanding and Applying the Health Benefits of Fasting. Obesity (Silver Spring). 2018 Feb;26(2):254-268. doi: 10.1002/oby.22065. Epub 2017 Oct 31. PMID 29086496
- [Background] Li C, Xing C, Zhang J, Zhao H, Shi W, He B. Eight-hour time-restricted feeding improves endocrine and metabolic profiles in women with anovulatory polycystic ovary syndrome. J Transl Med. 2021 Apr 13;19(1):148. doi: 10.1186/s12967-021-02817-2. PMID 33849562
- [Background] de Cabo R, Mattson MP. Effects of Intermittent Fasting on Health, Aging, and Disease. N Engl J Med. 2019 Dec 26;381(26):2541-2551. doi: 10.1056/NEJMra1905136. No abstract available. PMID 31881139
- [Background] Albosta M, Bakke J. Intermittent fasting: is there a role in the treatment of diabetes? A review of the literature and guide for primary care physicians. Clin Diabetes Endocrinol. 2021 Feb 3;7(1):3. doi: 10.1186/s40842-020-00116-1. PMID 33531076
- [Background] Zangeneh F, Salman Yazdi R, Naghizadeh MM, Abedinia N. Effect of Ramadan Fasting on Stress Neurohormones in Women with Polycystic Ovary Syndrome. J Family Reprod Health. 2015 Jun;9(2):51-7. PMID 26175759
- [Background] Pellegrini M, Cioffi I, Evangelista A, Ponzo V, Goitre I, Ciccone G, Ghigo E, Bo S. Effects of time-restricted feeding on body weight and metabolism. A systematic review and meta-analysis. Rev Endocr Metab Disord. 2020 Mar;21(1):17-33. doi: 10.1007/s11154-019-09524-w. PMID 31808043
- [Derived] Floyd R, Dyer A, Gibney J, Alawami F, Owens L, Phelan N, Rakovac A, Swan P, LeRoux CW, Behan LA, Duggan SN. Time-Restricted Eating to Improve Metabolic Abnormalities in Polycystic Ovarian Syndrome (TimeMAP). Clin Endocrinol (Oxf). 2026 Jan 14. doi: 10.1111/cen.70094. Online ahead of print. PMID 41532393
- See also: BDA The Association of UK Dieticians - Polycystic Ovary Syndrome (PCOS) Food Fact Sheet — https://www.bda.uk.com/resource/polycystic-ovary-syndrome-pcos-diet.html